CLINICAL TRIAL: NCT04126291
Title: Type 2 Diabetes Prevention Toolkit for Health-Care Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Principal Investigator, Jill Hamilton, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000060439
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Childhood Obesity
Keywords: education; health care professionals; type 2 diabetes; prevention
MeSH Terms: conditions — Pediatric Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The recruited group of health care professionals (HCPs) will answer a pre-questionnaire to collect demographic and practice data and ratings of perceived self-efficacy/confidence and knowledge in talking about weight-related issues. This pre-questionnaire only needs to be completed once. Participants will then be asked to watch each video. Immediately after watching each video, the participants will re-rate their perceived self-efficacy/confidence and knowledge to help elucidate outstanding educational gaps. For participants who consent to do a follow up questionnaire four-six months later, investigators will send an email link for HCPs to complete a satisfaction questionnaire and re-rate their perceived self-efficacy and knowledge to help elucidate outstanding educational gaps.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of whiteboard videos (Experimental): Participants will be provided an internet link via email to access the videos and questionnaires through REDCap (Research Electronic Data Capture), and responses will be tracked. Before viewing, participants will complete a pre-questionnaire to collect demographic and practice data and ratings of perceived self-efficacy/confidence and knowledge in talking about weight-related issues. This pre-questionnaire only needs to be completed once. Participants will then be asked to watch each video. Immediately after watching each video, participants will rate their perceived change in self-efficacy/ confidence and knowledge to help elucidate outstanding educational gaps. For those who consent to do a follow up questionnaire four-six months later, they will be sent an email link to complete a satisfaction questionnaire and rate their perceived self-efficacy/confidence and change in practice to help elucidate outstanding educational gaps.
  Interventions: Behavioral: Evaluation of whiteboard videos

INTERVENTIONS:
Behavioral: Evaluation of whiteboard videos — Participants will be provided an internet link via email to access the videos and questionnaires through REDCap (Research Electronic Data Capture), and responses will be tracked. Before viewing, participants will complete a pre-questionnaire to collect demographic and practice data and ratings of perceived self-efficacy/confidence and knowledge in talking about weight-related issues. This pre-questionnaire only needs to be completed once. Participants will then be asked to watch each video. Immediately after watching each video, participants will rate their perceived self-efficacy/confidence and knowledge to help elucidate outstanding educational gaps. For those who consent to do a follow up questionnaire four-six months later, they will be sent an email link to complete a satisfaction questionnaire and rate their perceived self-efficacy/confidence and change in practice to help elucidate outstanding educational gaps.

SUMMARY:
Tools are limited to help health care professionals talk about weight-related issues with their pediatric patients. The investigators have developed 6 whiteboard videos for health care professionals based on the 5As of Pediatric Obesity Management to address weight-related issues with pediatric patients and their families. This study aims to evaluate the videos using pre and post questionnaires. With the questionnaires, the investigators want to evaluate the content, quality (acceptability, engagement) and impact of patient-oriented educational videos on HCPs' self-efficacy/confidence and knowledge in regards to addressing weight-related issues with pediatric patients and their families using the 5A framework.

DETAILED DESCRIPTION:
Approximately one third of Canadian children and adolescents can be classified as having overweight or obesity. Health-care professionals (HCP), particularly primary care physicians, play a critical role in helping to address weight-related issues with patients and their families. A primary care-based obesity treatment model may be a practical means of treating obesity and helping to prevent Type 2 Diabetes and other co-morbidities. At the same time, obesity is not currently being addressed or managed in a consistent way across primary care settings, representing a significant gap in care. Furthermore, the extant literature indicates that HCPs feel ill-equipped to address obesity prevention and management, during childhood in particular. A lack of self-efficacy and training are recognized as two significant barriers to discussing weight with patients and their families. Other challenges for HCPs include the fear of damaging their relationship with patients and their families and the apprehension of triggering other issues such as eating disorders. For these reasons, effective educational materials are required for HCPs to promote healthy and helpful conversations about weight and risk of comorbidities. Research has shown that educational videos are an effective and engaging means to improve knowledge, confidence, and attitudes in HCPs and trainees. The investigators use The 5As of Pediatric Obesity Management as a framework for the creation of these educational videos. Preliminary evidence indicates that implementation of the 5As of Adult Obesity Management can increase communication amongst providers and patients in weight management. In 2013, experts from The Children's Hospital of Eastern Ontario (CHEO) partnered with CON to adapt this framework for use in a pediatric setting. It was designed as a step by step approach for busy primary care physicians who see childhood obesity in their practice. The Pediatric 5As presently exists as a downloadable booklet on the CON website. Although this resource is a helpful tool for HCPs, feedback from focus groups indicate that HCPs would like an expanded version with practical visuals of how a 5As framed encounter would occur in a busy office setting. The investigators have developed 6 videos to evaluate: Video #1: Weight Science 101, will present background information, including information on the factors driving body weight regulation. Video #2: A Word about BMI, will present background information on the advantages and disadvantages of using BMI. Video #3 ASK, reviews how to approach discussions about obesity with pediatric patients and their caregivers. Video #4: ASSESS, will review how to comprehensively assess children and youth with obesity. Video #5: ADVISE, AGREE, and ASSIST, will discuss the interventions for pediatric obesity management in the primary care setting, how to ensure patient engagement in the process, and how to sustain therapy. Our last video, Video #6: Putting it All Together, will summarize each of the 5As and how to use them as a comprehensive tool for pediatric obesity management.This study aims to evaluate the videos using pre and post questionnaires. With the questionnaires, the investigators want to evaluate the content, quality (acceptability, engagement) and impact of patient-oriented educational videos on HCPs' self-efficacy/confidence, knowledge, and change in practice in regards to addressing weight-related issues with pediatric patients and their families using the 5A framework.

ELIGIBILITY:
Inclusion Criteria:

* primary care family physicians
* pediatricians
* registered nurses
* nurse practitioners
* registered dietitians
* residents and fellows practicing in Canada.

Exclusion Criteria:

* inability to speak or read English fluently

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Change in self-efficacy/confidence related to pediatric obesity management | immediately after watching the video
  7 point likert scale where 1=no change or reduction in self-efficacy and 7= a great deal better
Change in knowledge | immediately after watching the video
  7 point likert scale where 1=no change or reduction in knowledge and 7= a great deal better

SECONDARY OUTCOMES:
Change in self-efficacy/confidence related to pediatric weight management | 4-6 months later
  A sliding scale from 0 to 100, where higher scores mean higher confidence. A mean change on the confidence scale between pre- and post-video.
Change in practice related to pediatric weight management | 4-6 months later
  7 point likert scale where 1=no change and 7=made all the difference in my practice

CONTACTS AND LOCATIONS:
Overall Officials: Jill K Hamilton, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The investigators plan to publish in a peer reviewed journal, as well as present at national and international conferences (Canadian Pediatric Endocrine Group, International Conference for Obesity and Canadian Pediatric Society )

REFERENCES:
- [Derived] Patel BP, Hadjiyannakis S, Clark L, Buchholz A, Noseworthy R, Bernard-Genest J, Walsh CM, McPherson AC, Strub J, Strom M, Hamilton JK. Evaluation of a Pediatric Obesity Management Toolkit for Health Care Professionals: A Quasi-Experimental Study. Int J Environ Res Public Health. 2021 Jul 16;18(14):7568. doi: 10.3390/ijerph18147568. PMID 34300020